CLINICAL TRIAL: NCT07311005
Title: THE EFFECT OF A NURSE-LED DIGITAL HEALTH EDUCATION PROGRAM ON BODY IMAGE SOCIAL PHYSIQUE ANXIETY AND MUSCLE DYSMORPHIA LEVELS IN YOUNG MEN WITH BIGOREXIA TENDENCIES: A RANDOMIZED CONTROLLED TRIAL
Brief Title: NURSE - LED DIGITAL EDUCATION AND BIGOREXIA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMU-BIGOREXIA-NURS-2025
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bigorexia; Muscle Dysmorphia; Wellness; Nurse-Led Digital Education
Keywords: Muscle Dysmorphia; Male Body İmage; Health Behavior; Bigorexia; Wellness; Nursing
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Digital Education
- Control Group (No Intervention)

INTERVENTIONS:
Other: Digital Education — In the study, the intervention group will receive a digital-based "Healthy Lifestyle Education for Bigorexia" consisting of 12 sessions. Each session will be conducted as an interactive module lasting approximately 60 minutes. The education will cover topics including balanced nutrition, regular physical activity, development of a healthy body image, and strategies for coping with social physique anxiety.
  The educational materials will consist of video presentations, brief reading materials, and interactive exercises. Participants' questions throughout the training will be addressed via online discussion platforms. At the end of the study, the scale-based assessments will be re-administered.
  Arms: Intervention Group

SUMMARY:
In recent years, the desire to achieve a muscular body appearance has been increasingly observed among young men, and this situation may lead to unhealthy behaviors and psychological problems in some individuals. Bigorexia, also referred to as muscle dysmorphia, is considered a significant condition within body image disorders and is characterized by a persistent and unrealistic perception of not being sufficiently muscular.

Young men with tendencies toward bigorexia may experience negative body image, feel anxiety related to their physical appearance in social settings, and consequently suffer a decline in their quality of daily life. This phenomenon, which can lead to serious psychological, physical, and social problems, plays an important role in the lives of men. The present study aims to examine the effects of a 12-week digital-based education program provided to young men with bigorexia tendencies on body image, social physique anxiety, and levels of bigorexia.

In this research, the effects of a digital-based health education program developed for young men with bigorexia tendencies will be investigated. The study will be conducted using a randomized controlled experimental design, and the impact of the digital health education on participants' body image, social physique anxiety, and bigorexia levels will be evaluated. It is expected that the findings will provide evidence-based data to support the development of healthy lifestyle behaviors among young men, strengthen positive body image, and reduce the risk of bigorexia. Additionally, demonstrating the effectiveness of digital-based educational interventions is anticipated to introduce an innovative approach to public health nursing practice.

ELIGIBILITY:
Inclusion Criteria:

Being between 18-30 years of age

Being male

Actively attending a gym/fitness center

Providing voluntary informed consent to participate in the study

Scoring 39 or above on the Bigorexia Scale

Exclusion Criteria:

Being female

Having a communication impairment

Not attending the education program for more than two weeks

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 18- 30 years old man
Enrollment: 68 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pre-test-post-test education score difference | 8 month

CONTACTS AND LOCATIONS:
Locations (1):
- EMU, Mersin, Mağusa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No